CLINICAL TRIAL: NCT02166554
Title: The Efficacy and Safety of a New Cross-linked Hyaluronan Hydrogel in the Reduction of Postsurgical Adhesions After Laparoscopic Gynecological Surgery: a Randomized Controlled Trial
Brief Title: The Efficacy and Safety Study of a New Cross-linked Hyaluronan Hydrogel in the Reduction of Postsurgical Peritoneal Adhesions
Acronym: BAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioRegen Biomedical (CHangzhou) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FNL-2011-05
Record Dates: First submitted 2014-06-13; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Myomas; Ovary Cysts; Endometriotic Cysts; Adhesions
Keywords: Adhesions; Hyaluronan; Gynaecological surgery; Clinical outcomes
MeSH Terms: conditions — Myoma; Tissue Adhesions | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Placebo Comparator): Standard of care for post-operative adhesion prevention included irrigation of tissues and lavage of all fluids with saline placebo following surgery
  Interventions: Other: Saline
- Cross-linked Hyaluronan Hydrogel Arm (Experimental): HyaRegen
  Interventions: Device: Cross-linked Hyaluronan Hydrogel

INTERVENTIONS:
Other: Saline — On the day of initial surgery
  Arms: Control Arm
Device: Cross-linked Hyaluronan Hydrogel — On the day of the initial surgery
  Other Names: HyaRegen; Self Cross-linked Hyaluronan Gel
  Arms: Cross-linked Hyaluronan Hydrogel Arm

SUMMARY:
The purpose of this study was to determine whether the new crosslinked hyaluronan hydrogel was safe to use, and was effective for the prevention/reduction of adhesion formation following gynecological surgery

DETAILED DESCRIPTION:
Postsurgical adhesions are a common medical complication of gynecologic and pelvic surgeries, and are frequently associated with chronic or recurrent pelvic pain, intestinal obstruction and infertility. This randomized, controlled, multicenter, clinical study was designed to evaluate the safety and performance of the new crosslinked hyaluronan hydrogel versus the standard of care for the reduction of postoperative adhesions in subjects undergoing laparoscopic surgeries. Subjects were scheduled to return at 9 weeks after the initial surgical procedure. At that time, a second-look laparoscopy was performed for postsurgical adhesion assessment. Adhesions were graded using a modified American Fertility Society (mAFS) scoring system.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Aged 18-45 years.
* Been scheduled for removal of myomas, ovary cysts, endometriotic cysts or adhesions.
* Been willing to comply with all aspects of the treatment and evaluation schedule.
* Agreed to a second-look laparoscopic procedure to assess and lyse any adhesions formed at 9 weeks following the primary surgery.
* Provided voluntary written informed consent.

Exclusion Criteria:

* Acute or severe infection.
* Autoimmune diseases such as diabetes etc.
* Abnormal liver/renal and cardiovascular function
* Abnormal blood coagulation
* Medical histories of peripheral vascular disease, alcohol or drug abuse, and mental illness.
* Known or suspected intolerance or hypersensitivity to hyaluronan or its derivatives.
* Concurrent use of systemic antiinflammatory drugs.
* Clinical evidence of cancer.
* Use of anticoagulant, fibrin glue, other thrombogenic agents, or any other anti-adhesion agent during the procedure.
* Concurrent peritoneal grafting or tubal implantation.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2011-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The adhesion incidence under moderate/severe category | 9 weeks following primary laparoscopic gynecological surgery
  The patient percentage with modified American Fertility Society (mAFS) score (ovaries and tubes) more than 4 points.

SECONDARY OUTCOMES:
modified American Fertility Society (mAFS) score | 9 weeks following primary laparoscopic gynecological surgery
  modified American Fertility Society (mAFS) score of ovaries/tubes
Adhesion extent | 9 weeks following primary laparoscopic gynecological surgery
  Adhesion extent of ovaries/tubes
Adhesion severity | 9 weeks following primary laparoscopic gynecological surgery
  Adhesion severity of ovaries/tubes
The adhesion incidence under moderate/severe category | 9 weeks following primary laparoscopic gynecological surgery
  The patient percentage with modified American Fertility Society (mAFS) score (throughout abdominopelvic cavity) more than 4 points.
modified American Fertility Society (mAFS) score | 9 weeks following primary laparoscopic gynecological surgery
  modified American Fertility Society (mAFS) score (throughout abdominopelvic cavity)
Adhesion extent | 9 weeks following primary laparoscopic gynecological surgery
  Adhesion extent (throughout abdominopelvic cavity)
Adhesion severity | 9 weeks following primary laparoscopic gynecological surgery
  Adhesion severity (throughout abdominopelvic cavity)
Adverse events | Up to 9 weeks
  Safety evaluation was based on clinical laboratory tests, the type and severity of adverse events recorded throughout the study, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Zhang, MD, PhD, Principal Investigator — Beijing Chao Yang Hospital
Locations (7):
- China (7):
  - Beijing Chao-Yang Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Xiangya Hospital, Changsha, Hunan
  - Qilu Hospital, Jinan, Shandong

REFERENCES:
- [Derived] Liu C, Lu Q, Zhang Z, Xue M, Zhang Y, Zhang Y, Wang H, Li H, Zhou Y, Zhang Z, Li W; HyaRegen Adhesion Study Group. A Randomized Controlled Trial on the Efficacy and Safety of a New Crosslinked Hyaluronan Gel in Reducing Adhesions after Gynecologic Laparoscopic Surgeries. J Minim Invasive Gynecol. 2015 Jul-Aug;22(5):853-63. doi: 10.1016/j.jmig.2015.04.011. Epub 2015 Apr 20. PMID 25906706